CLINICAL TRIAL: NCT03561350
Title: Detect Microsatellite Instability Status in Blood Sample of Advanced Colorectal Cancer Patients by Next-Generation Sequencing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Other Study IDs: MISC-MSI
Record Dates: First submitted 2018-05-25; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Neoplasms
Keywords: Microsatellite Instability; Circulating Tumor DNA; Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Microsatellite Instability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample of advanced colorectal cancer patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The method to analyze the microsatellite instability (MSI) status by next-generation sequencing (NGS) has been established to assess the deficiency of DNA mismatch repair (MMR) system. The aim of our study is to evaluate the feasibility and reliability of this NGS method by testing the circulating tumor DNA (ctDNA) in blood sample of advanced colorectal cancer patients. If the result is positive, the MSI status could be easily learned without the acquisition of tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* a biopsy proven histological diagnosis of colorectal carcinoma
* MSI status of tissue sample known by IHC or PCR method
* willing to participate and informed consent signed

Exclusion Criteria:

* history of other malignant tumors
* patients with inflammatory bowel disease
* patients with familial adenomatous polyposis
* patients treated by surgery or adjuvant treatment
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in Shanghai Minimally Invasive Surgery Center
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-09-28 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
MSI status in blood sample | through study completion, an average of 1 year
  ctDNA and leucocyte are extracted from blood sample for MSI detection by ColonCore NGS panel (Burning Rock, Guangzhou, China). There are three types of MSI status, MSI-H, MSI-L and MSS.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Minimally Invasive Surgery Canter, Ruijin hospital, Shanghai, Shanghai Municipality, China